CLINICAL TRIAL: NCT00713076
Title: Wettability of Contact Lenses With a Multi-Purpose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-07-18
Record Dates: First submitted 2008-06-18; First posted 2008-07-11 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2008-07

CONDITIONS: Vision
Keywords: multi-purpose solution; contact lens wearers; Contact lense wearers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Polyquaternium-preserved Multi-purpose solution
  Interventions: Other: Polyquaternium-preserved Multi-purpose Lens Cleaning Solution 109182

INTERVENTIONS:
Other: Polyquaternium-preserved Multi-purpose Lens Cleaning Solution 109182 — Lens Cleaning Solution Formulation Identification Number 109182

SUMMARY:
Measure wettability of hydrogel and silicone hydrogel contact lenses presoaked in a Multi-Purpose Solution.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal eyes who have successfully worn contact lenses on a daily basis for at least two weeks prior to the study.
* Must be wearing lenses a minimum of eight hours a day
* Vision must be correctable to 20/30 (snellen) or better in each eye at a distance with soft contact lenses
* Use no topical ocular OTC or prescribed ocular medication

Exclusion Criteria:

* Subjects with current lid or conjunctival infections, abnormalities, inflammation, abnormal corneal opacities, significant lenticular inclusions, iritis, ocular disease or condition, corneal surgery, cataract surgery, intraocular lens implants, or glaucoma filtering surgery.
* Subjects using systemic medications, upper respiratory infections or colds, history of seasonal allergies with significant ocular side effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Lens Wettability - ex-vivo wetting angle | From baseline

SECONDARY OUTCOMES:
Slit-lamp findings Corrected visual acuity (snellen) Adverse events | From baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Study Locations, Fort Worth, Texas, United States